CLINICAL TRIAL: NCT07219797
Title: Study of Monochromatic X-ray Mammography System
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Imagine Scientific, Inc. (Industry)
Collaborators: Duke Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: Pro00115443
Record Dates: First submitted 2025-09-11; First posted 2025-10-22 (Actual); Last update posted 2025-10-22 (Actual); Status verified 2025-10

CONDITIONS: Breast Imaging; Breast Cancer
Keywords: Mammography
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Test device vs standard of care (Experimental): Demonstrate that a 2-D monochromatic x-ray mammography system can produce mammographic images using lower radiation dose, yet not inferior to conventional mammography.
  Interventions: Device: 2-D Monochromatic X-ray Mammography System

INTERVENTIONS:
Device: 2-D Monochromatic X-ray Mammography System — Monochromatic x-ray mammography system produces superior images as compared to conventional 2-D and 3-D mammography while using a lower radiation dose.

SUMMARY:
A research study to find out if an investigational mammography machine is effective in producing high-quality images using a lower radiation dose than traditional mammography.

DETAILED DESCRIPTION:
Prospective, single-arm, non-blinded, comparative/observational study.

Phase 1: Verify operation of monochromatic system and optimize the monochromatic energies and exposure times for a range of breast thicknesses.

Phase 2: Test the performance of the monochromatic system in comparison to traditional 2-D mammography for a range of clinical/imaging scenarios.

Phase 3: Test the performance of the monochromatic system using reduced breast compression.

ELIGIBILITY:
Inclusion Criteria:

* Female
* 40 yrs of age or older
* Capable of giving informed consent
* Prior history of mammography

Exclusion Criteria:

* Pregnancy
* History of breast cancer surgery, including lumpectomy or mastectomy
* Currently undergoing treatment for breast cancer
* Previous breast augmentations

Min Age: 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Noninferiority of a 2-D monochromatic X-ray mammography system compared to conventional mammography | Enrollment to end of visit 1 (or up to 7 days following visit 1, if needed)
  Demonstrate that a 2-D monochromatic X-ray mammography system can produce mammographic images using lower radiation dose (at least 20% less than conventional mammography), yet, not inferior to conventional mammography. [Likert scale 1-3. Higher score is a better outcome]

SECONDARY OUTCOMES:
Relevant pathologies identified by monochromatic-based x-ray as compared to conventional mammography | End of visit 1 (or up to 7 days following visit 1, if needed)
  Assess ability of monochromatic-based X-ray mammography to identify relevant pathologies in subjects with dense breast issue (BI-RADS density categories C and D) otherwise not detected in scans produced with conventional mammography. [Likert scale 1-3. Higher score is a better outcome]
Lower breast compression with monochromatic-based x-ray mammography | Enrollment to end of visit 1 (or up to 7 days following visit 1, if needed)
  Assess ability of monochromatic-based x-ray mammography to produce quality images with lower breast compression. [Likert scale 1-3. Higher score is a better outcome]
Quality of images produced by monochromatic-based x-ray mammography at lower radiation dose. | Enrollment to end of visit 1 (or up to 7 days following visit 1, if needed)
  Demonstrate ability of monochromatic-based mammography to produce quality images at radiation doses below maximum FDA-approved radiation dose. [Likert scale 1-3. Higher score is a better outcome]
Patient satisfaction with monochromatic x-ray mammography system | Enrollment to end of visit 1 (or up to 7 days following visit 1, if needed)
  Assess patient satisfaction with monochromatic x-ray mammography system. [Likert scale 1-5. Higher score is a better outcome.]

CONTACTS AND LOCATIONS:
Overall Officials: Lars Grimm, MD, Principal Investigator — Duke Health
Locations (1):
- Duke Cancer Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
Data is confidential and proprietary. Sponsor permission is required to share data.